CLINICAL TRIAL: NCT06886282
Title: Spatial RadiomIcs and TRanscriptomics to the DIscovery of the Cross-link Between Colon Cancer and ChrOnic Kidney Disease
Acronym: SIRIO
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Principal Investigator, Antonella Petrillo, National Cancer Institute, Naples, National Cancer Institute, Naples
Other Study IDs: PNRR-MCNT1-2023-12378005
Record Dates: First submitted 2025-03-12; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Cancer (CRC)
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The incidence of colorectal cancer (CRC) is higher in patients with chronic kidney disease (CKD) compared to general population. Causal factors have not been clarified so far, although some hypothesis could be formulated. Tumor microenvironment (TME) impacts cancer progression and is influenced by different chronic diseases associated with systemic inflammation. In our study, we aim to address this relevant issue by an in-deep characterization of TME in CKD patients with CRC undergoing surgery. This will provide genes expression directly on tumor tissues.

Our network includes three high national relevance hospitals (INT IRCCS Pascale, AOU Vanvitelli and AOU Brotzu) and a Genetic Research Institute (Biogem Scarl). We will recruit two comparing groups of CRC patients eligible for surgical cancer resection: 1. Patients with I-II stage CRC alone, and 2. Patients with I-II stage CRC and CKD. Anthropological, clinical and laboratory tests data will be collected and organized in a database for epidemiological and descriptive analysis of the enrolled cohorts. Patients will be matched by age, gender and cancer stage and will be stratified by the estimated renal function (application of BSA eGFR formula by Janovitz T et al, J Clin Oncol, 2017). Patients will undergo preoperative high resolution abdominal MRI for high throughput accurate macroscopic assessment of TME by radiomic approach. During surgery, tumor tissue samples will be collected and promptly frozen at -80°C for subsequent analysis. CRC tissue samples will be analyzed combining spatially resolved and single-cell transcriptomic approach, providing a sensitive and unbiased lens for identifying the key mechanisms of the interplay between CRC and immune context, preserving their tissue architecture. Our study involves the usage of Visium Cytassist Spatial Gene Expression, a powerful tool based on in situ capturing methods, providing the whole transcriptome information from tissue sections.

Data collected by radiomics and tissue transcriptomics will undergo integrated analysis by a bioinformatic approach based on computational methods. TME will be macroscopically characterized on tumor images to map specific tissue areas of interest.

By spatial tumor sections analysis, initial segregation of non-malignant TME cells from malignant ones will be performed and then the identification of differentially expressed genes and pathways between the two groups of patients will be finalized.

These methodologies will allow the full characterization of CRC environment and will highlight possible differences between groups in TME macroscopic imaging features and gene expression. This will permit the discovery of possible specific tumor imaging-detected patterns and the associated molecular pathways specially promoted or deregulated in CKD patients with CRC. These evidences will enhance the value of possible prognostic parameters and the identification of early biomarkers of CRC and future development of targeted therapies. In the era of precision medicine, these goals appear relevant to address the increasing cost and social impact of both CRC and CKD.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Life expectancy greater than 3 months **
* Histopathological diagnosis of colorectal cancer stage I or II according to the TNM (Tumor, Node, Metastasis) classification
* Patients with tumors classified as T1-T3, N0, M0 (stage I-II) eligible for surgery
* Ability to understand and sign the informed consent
* Clinically stable patients with no significant changes in renal function or disease management in the weeks prior to enrollment **

For the non-CKD group

• Adequate liver, renal and bone marrow function (adequate levels of hemoglobin, platelets, creatinine and bilirubin)

For the CKD group

* Confirmed diagnosis of chronic kidney disease according to the KDIGO (Kidney Disease: Improving Global Outcomes) guidelines defined by a duration of at least three months with structural or functional abnormalities of the kidneys
* BSA (Body Surface Area Area) eGFR≤60 ml/min/1.73 m2

Exclusion Criteria:

* Recent episodes of acute renal failure
* Kidney transplant, autoimmune diseases; inflammatory bowel diseases; other than oncological or oncohematological diseases of CRC
* Recent therapies with steroids/immunosuppressants and cardiovascular events (within 3 months of enrollment)
* History of serious allergic reactions to iodinated contrast agents or gadolinium-based contrast agents
* Recent or planned invasive or surgical treatments that could interfere with the study (within 3 months of enrollment)
* Psychiatric disorders that could impair the patient's ability to follow study procedures or provide informed consent
* Other types of concomitant or previous tumors in the previous 5 years of enrollment
* Pregnant or breastfeeding women. Pregnancy status will be ascertained before enrollment by measuring Beta-hCG in urine (Pregnancy Test or urinary beta-HCG) or in blood (plasma beta-hCG).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Two groups of CRC patients who are candidates for endoscopic or surgical resection of the cancer will be recruited:
  1. Patients with stage I-II CRC without CKD
  2. Patients with stage I-II CRC with CKD
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-11-05 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Identification of specific biomarkers by transcriptomic study | through study completion, an average of 2 years
  Identification of specific biomarkers by transcriptomic study among patients with stage I-II CRC and CKD and patients with stage I-II CRC without CKD undergoing endoscopic or surgical tumor removal.

SECONDARY OUTCOMES:
Identification of specific biomarkers by radiomics study | through study completion, an average of 2 years
  Identification of specific biomarkers by Radiomics study on baseline radiological examinations performed before endoscopic or surgical resection, among patients with stage I-II CRC and CKD and patients with stage I-II CRC without CKD.

CONTACTS AND LOCATIONS:
Locations (1):
- Radiology Division, Naples, Italy